CLINICAL TRIAL: NCT05508191
Title: Microneedling Versus Fractional CO₂ Laser Resurfacing for Skin Rejuvenation With Adipose-derived Mesenchymal Stem Cells Secretome: a Single-blind, Randomized Clinical Trial
Brief Title: Microneedle Versus Fractional CO₂ Laser for Skin Aging Treatment With Stem Cell Secretome in Indonesian Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shannaz Nadia Yusharyahya (Other)
Collaborators: PT. Kimia Farma (Persero) Tbk (Industry); Ministry of Education, Culture, Research, and Technology, Republic of Indonesia (Unknown)
Responsible Party: Sponsor-Investigator, Shannaz Nadia Yusharyahya, Head of Geriatric Dermatology Division, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia-dr. Cipto Mangunkusumo Hospital, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-08-0682
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Skin Aging; Transepidermal Water Loss
Keywords: Adipose-derived mesenchymal stem cells; Fractional CO₂ laser; Microneedling; Secretome; Skin rejuvenation

STUDY DESIGN:
Intervention Model Description: Each participant will receive fractional CO₂ laser treatment on one side of the face and microneedle treatment on the other half. The allocation of which side receive a particular treatment will be determined by a computer programme.
Who Masked: Outcomes Assessor
Masking Description: The investigator (who evaluated the skin aging status, or the outcomes assessor) will be blinded to the treatment allocation until the end of data collection. We cannot perform the masking to the participants as they will surely aware which side of their face receive microneedle or fractional CO₂ laser, even though they are required to close their eyes during treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secretome + Fractional CO₂ Laser (Experimental): This clinical study uses a 4-fold concentrate of ADMSCs secretome developed by PT. Kimia Farma (Persero), Tbk. The secretome is extracted from stem cell line filtered through syringe with pore size of 0.22 µm to eliminate the debris, then concentrated with CorningⓇ Spin-XⓇ UF 500 µL centrifugator. Stabilization analysis is performed before utilization. As for fractional CO₂ laser, AMIⓇ device is used with this following settings: 15 mJ energy, 900 µs pulse duration, density level 15, and depth level 2.
  Interventions: Device: Fractional CO₂ Laser
- Secretome + Microneedle (Experimental): This clinical study uses a 4-fold concentrate of ADMSCs secretome developed by PT. Kimia Farma (Persero), Tbk. The secretome is extracted from stem cell line filtered through syringe with pore size of 0.22 µm to eliminate the debris, then concentrated with CorningⓇ Spin-XⓇ UF 500 µL centrifugator. Stabilization analysis is performed before utilization. As for microneedle, DrPenⓇ dermapen is used in this following direction and order: vertical, horizontal, and diagonal, with the depth of 150 µm.
  Interventions: Device: Microneedle

INTERVENTIONS:
Device: Fractional CO₂ Laser — Prior to the treatment, each participant will be evaluated for their initial skin status, followed by daily priming with 0.05% retinoic acid cream, applied topically at night for two weeks. At second week, the participants will undergo facial skin anesthesia utilizing 2.5% lidocaine+2.5% prilocaine cream for 30 minutes. Half of the face will be irradiated with AMIⓇ fractional CO₂ laser according to the instrument manual for 20 minutes, succeeded by the topical administration of 1.5 mL 4-fold concentrated ADMSCs secretome. The participants are all instructed not to: (1) wash their face for the next 4 hours; (2) apply sunscreen for the next 1 day; and (3) apply retinoic acid cream for the next 3 days. After the restriction, they should use the mentioned products on daily basis until the next appointment when the protocol is repeated (fourth week). At sixth week, the final skin condition is reevaluated with the same tools, along with the additional variables.
  Arms: Secretome + Fractional CO₂ Laser
Device: Microneedle — Prior to the treatment, each participant will be evaluated for their initial skin status, followed by daily priming with 0.05% retinoic acid cream, applied topically at night for two weeks. At second week, the participants will undergo facial skin anesthesia utilizing 2.5% lidocaine+2.5% prilocaine cream for 30 minutes. The other half of the face will be treated with DrPenⓇ dermapen according to the instrument manual for 20 minutes, succeeded by the topical administration of 1.5 mL 4-fold concentrated ADMSCs secretome. The participants are all instructed not to: (1) wash their face for the next 4 hours; (2) apply sunscreen for the next 1 day; and (3) apply retinoic acid cream for the next 3 days. After the restriction, they should use the mentioned products on daily basis until the next appointment when the protocol is repeated (fourth week). At sixth week, the final skin condition is reevaluated with the same tools, along with the additional variables.
  Arms: Secretome + Microneedle

SUMMARY:
Evidences regarding the effectiveness of adipose-derived mesenchymal stem cells (ADMSCs) secretome to alleviate skin aging have been extensively available, yet no studies hitherto directly investigated the best administration technique for such purpose. The objective of this study is to compare microneedling and fractional CO₂ laser methods in administrating ADMSCs secretome for facial skin rejuvenation of Indonesian adult women.

DETAILED DESCRIPTION:
A single-blind, randomized clinical trial will be conducted upon thirty females (aged 35-59 years old) presented with signs of generalized facial cutaneous senescence. Their initial skin status will be evaluated utilizing dermoscopy photoaging scale (DPAS) and Janus-3® skin analyzer, along with skin capacitance using the Corneometer® and transepidermal water loss using the Tewameter®, followed by daily priming with 0.05% retinoic acid for two consecutive weeks. At second and fourth week, the participants are subjected to microneedle and fractional CO₂ laser according to the respective protocol in split-face fashion, which the randomization will be determined by a computer programme. Succeeding the treatment, four-fold concentrated ADMSCs secretome will be administered topically to the both sides of face. The final skin condition will ultimately be recorded at the sixth week, along with their satisfaction and convenience degree, the adverse events experienced during the trial, and subjective preference to the treatment. Appropriate statistical analyses will subsequently be performed at the significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 35-59 years
* Generalized wrinkles on the face
* Consent for the 2-month clinical trial (4 times of follow-up with 2 weeks interval)

Exclusion Criteria:

* Prior history of hypertrophic scars or keloid formation
* Prior history of allergy to topical anesthetic and/or retinoic acid cream
* Prior history of autoimmune disorders (e.g. systemic lupus erythematosus, rheumatoid arthritis, etc.)
* Prior history of malignancies
* Prior utilization of skincare products for the past 6 months
* Currently under long-term immunosupressants medication (e.g. corticosteroids, biologic agents, cytostatics, etc.)

Drop-out Criteria:

* Pass away during the clinical trial
* Refrain from the clinical trial before the trial completion
* Absent for more than two days from the scheduled appointment
* Suffer from coronavirus disease 2019 (COVID-19) at any time during the trial
* Experience major adverse event(s) caused by topical products or treatments given in the clinical trial (e.g. allergic drug eruption or contact dermatitis). The participants will receive appropriate management if such event occurs.

Ages: 35 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Skin aging changes evaluated by dermoscopy photoaging scale (DPAS) | Week 0 (baseline), week 2 before intervention, week 4 before intervention, week 6 (end of trial)
  A thorough evaluation using dermoscope upon 11 parameters of skin aging (yellowish papules, solar elastosis, skin atrophy, lentigo, hypopigmented and hyperpigmented macules, telangiectasia, actinic keratosis, senile comedones, superficial wrinkles, deep wrinkles, and criss-cross wrinkles) observed on 4 locations (forehead, periorbita, zygoma, and mandible). Each finding on each location has a value of 1, so the maximum possible total score is 44.
  *This is a numeric variable.
Skin aging changes evaluated by Janus-3Ⓡ skin analyzer | Week 0 (baseline), week 2 before intervention, week 4 before intervention, week 6 (end of trial)
  A comprehensive evaluation using Janus-3Ⓡ skin analyzer upon 4 parameters of skin aging (wrinkle, pore size, pigmentation, and sebum) observed on the same location for each assessment. Each finding is expressed as percentage (%).
  *This is a numeric variable.
Skin capacitance evaluated by the CorneometerⓇ | Week 0 (baseline), week 2 before intervention, week 4 before intervention, week 6 (end of trial)
  Total water content in the stratum corneum of the skin, reported in microsiemens.
  *This is a numeric variable.
Transepidermal water loss evaluated by the TewameterⓇ | Week 0 (baseline), week 2 before intervention, week 4 before intervention, week 6 (end of trial)
  Water evaporation rate in a given area of skin, reported in gram/m²/hour.
  *This is a numeric variable.

SECONDARY OUTCOMES:
Likert scale for the satisfaction degree | Week 6 (end of trial)
  An interval of 0 (extremely unsatisfied) to 10 (extremely satisfied) for determination of the participants' satisfaction upon both treatments (microneedle and fractional CO₂ laser).
  *This is a numeric variable.
Visual analog scale (VAS) of pain for the convenience degree | Week 6 (end of trial)
  An interval of 0 (no pain whatsoever) to 10 (the most extreme pain possible) for determination of the participants' convenience during the trial with both treatments (microneedle and fractional CO₂ laser).
  *This is a numeric variable.
Number of adverse events experienced during the clinical trial | Week 2 thirty minutes after intervention, week 4 thirty minutes after intervention, week 6 (end of trial)
  Side effects experienced by the participants following the application of topical products (facial wash, sunscreen, anesthetic cream, and retinoic acid cream) and procedures (microneedle and fractional CO₂ laser), such as erythema, warmth, itch, burning sensation, edema, peeled skin, and/or no adverse events, reported in frequency of each event. Each participant will be contacted one day after each treatment for side effect evaluation. They can also report any events experienced to the investigator at any time during the trial.
  *This is a categorical variable.
Subjective preference to treatment | Week 6 (end of trial)
  Preference of each subject towards a particular treatment (microneedling or fractional CO2 laser) based on their experience during the trial
  *This is a categorical variable

CONTACTS AND LOCATIONS:
Overall Officials: Endi Novianto, MD, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Irma Bernadette, MD, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Lili Legiawati, MD, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Noer Kamila, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No